CLINICAL TRIAL: NCT03352609
Title: Accelerated Repetitive Transcranial Magnetic Stimulation (rTMS) of the Dorsolateral Prefrontal Cortex for the Reduction of Craving in Nicotine Dependent Individuals
Brief Title: Accelerated rTMS for the Reduction of Nicotine Craving
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator completing residency program and leaving for a new job
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, David Friedrich, Resident Physician, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00070449
Record Dates: First submitted 2017-11-08; First posted 2017-11-24 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Nicotine Use Disorder; Nicotine Dependence
Keywords: TMS; rTMS; Transcranial Magnetic Stimulation; Smoking; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized double blind control using a sham rTMS system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active rTMS (Experimental): 5 sessions of rTMS delivered with MagPro (MagVenture) double blind rTMS system delivered at 110% of resting motor threshold with 3000 pulses of 10hz stimulation (5s on, 10s off) per session.
  Interventions: Device: Active rTMS with MagVenture MagPro double blind rTMS system
- Sham (Sham Comparator): 5 session of sham rTMS delivered with Magpro (MagVenture) double blind rTMS system to mimic active intervention.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS with MagVenture MagPro double blind rTMS system — 5 sessions of rTMS delivered with MagPro (MagVenture) double blind rTMS system delivered at 110% of resting motor threshold with 3000 pulses of 10hz stimulation (5s on, 10s off) per session.
  Arms: Active rTMS
Device: Sham rTMS — Double blind MagPro system delivers sham condition by mimicking rTMS sound and delivering skin stimulus via TENS pads
  Arms: Sham

SUMMARY:
The purpose if this study is to determine if five treatments of repetitive transcranial magnetic stimulation (rTMS) can reduce craving for cigarettes in smokers. rTMS uses magnetic pulses to stimulate the brain and is currently approved for the treatment of major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient Adults aged 18-70
* Cigarette Smokers smoking at least 1 pack (20 cigarettes a day) with current smoking status confirmed by exhaled CO reading of >10ppm day of visit.
* Ability to provide informed consent

Exclusion Criteria

* Current treatment with varenicline or bupropion
* Currently making a smoking quit attempt (not currently smoking).
* Current treatment with an antidepressant, anti-convulsant, anxiolytic, antipsychotic or mood stabilizer.
* Current episode of major depression determined by MINI interview.
* Current or past history of schizophrenia, schizoaffective disorder, anorexia nervosa, bulimia or bipolar disorder as determined by MINI.
* Current daily consumption of alcohol or current alcohol use disorder.
* Current substance use disorder except for nicotine or cannabis use disorder.
* Currently pregnant or lactating.
* Contraindications to rTMS including history of seizure, metal implanted above the neck, pacemaker or any brain lesion.
* Unstable medical conditions
* Suicidal ideation or history of suicide attempt within the last six months.
* Inability or unwillingness of subject or legal guardian/representative to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Friedrich, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS | Sham
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Tolerability Measured by Percent of Participants Completing the rTMS Course
Description: Percent of participants completing the 5 session rTMS course. Hypothesize >75% of participants will complete the 5 treatments.
Time Frame: 1 day (single visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Active rTMS | Sham
Number analyzed (Participants) | 2 | 3
Participants | 2 | 3

2. Primary Outcome: Decrease in Cue Induced Nicotine Craving
Description: Nicotine craving evaluated using Questionnaire on Smoking Urges- Brief (QSU-B) questions modified to a 0-100 analog rating. Higher scores meaning a higher level of craving.
Time Frame: During the one day visit
Measure: Mean (Full Range); unit: Percent change on craving scale
Arm/Group | Active rTMS | Sham
Number analyzed (Participants) | 2 | 3
Percent change on craving scale | -4.65 [-10 to 0.7] | -7.6 [-21.3 to 3.3]

3. Secondary Outcome: Reduce in Self Reported Smoking
Description: An exploratory outcome will be the determination if participants receiving active rTMS report decreased levels of smoking 1 week and 2 weeks after rTMS course.
Time Frame: 1 week and 2 weeks after rTMS
Population: Participants did not return follow up phone call
Arm/Group | Active rTMS | Sham
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Single visit of approximately 6 hours
Arm/Group | Active rTMS | Sham
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/2 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active rTMS (N=2) | Sham (N=3)
Slight scalp discomfort (Skin and subcutaneous tissue disorders) | 1 | 0 — Immediately resolved
Mild Nausea (General disorders) | 0 | 1 — transient, self resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT03352609/Prot_SAP_000.pdf